CLINICAL TRIAL: NCT05765552
Title: Effects Of Dual-Task Training On Balance, Fear Of Falling,Cognitive Functions, Dual-Task Performance, Depression And Quality Of Life In Individuals With Alzheimer
Brief Title: Effects of Dual-Task Training In Individuals With Alzheimer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Mehmet Ozkeskin, Asisstant Professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOzkeskin874
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer; Fear of falling; Dual-task; Balance; Cognition
MeSH Terms: conditions — Alzheimer Disease | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Participants in control group will receive an exercise program consisted of upper and lower range of motion exercises.The exercises will be started as 8-10 repetitions and 1 set and the number of sets will be increased according to the progression of the patient. Exercises will be applied for 8 weeks, 2 days a week, each session will last for 30 minutes.
  Interventions: Other: Control Group
- Dual-Task Training Group (Experimental): Participants in the dual-task training group will receive exercises involving both motor and cognitive functions.Dual-task training sessions will begin with 10 minutes of stretching and proceed with 20 minutes of motor-cognitive dual-task exercises (counting backwards from 30 on double stance, naming the months and singing when standing on soft surfaces, finding words that starts with a given letter etc.) and sessions will end with 10 minutes of cooling.Exercises will be applied for 8 weeks 2 days a week each session will last for 30 minutes.
  Interventions: Other: Dual-Task Training

INTERVENTIONS:
Other: Dual-Task Training — Motor-cognitive dual-task exercises will be applied for 2 days a week for 8 weeks.Sessions will last for 30 minutes.
  Arms: Dual-Task Training Group
Other: Control Group — Upper and lower extremity range of motion exercises will be applied for 8-10 repetitions for 1 set 2 times a week for 8 weeks.
  Arms: Control Group

SUMMARY:
The purpose of this study is to investigate the effects of dual-task training on balance, fear of falling, cognitive functions, dual-task performance, depression and quality of life in individuals with Alzheimer.

DETAILED DESCRIPTION:
Eligible participants will be randomized to control or dual-task training group.Control group will receive conventional therapy generally consisted of lower and upper range of motion exercises for 30 minutes 2 times a week for 8 weeks.Dual-task training group will receive exercises involving motor-cognitive dual-task exercises for 30 minutes 2 times a week for 8 weeks.Each participant will be assessed before and after the 8 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* having been diagnosed with mild or moderate Alzheimer's disease
* able to walk with or without assistance
* having sufficient visual and auditory ability to perform the cognitive tests
* being fit to perform physical exercises
* being able to participate in proposed interventions and assessments

Exclusion Criteria:

* having a neurological disorder other than Alzheimer
* having any musculoskeletal problems that can affect balance
* having any contraindication to exercise
* functional limitation or sensory impairment that may affect performance
* major depression

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Timed Up And Go(TUG) | eight weeks
  It is a frequently used test that evaluates functional mobility and dynamic balance. At the beginning of the test, individuals sit in a chair. A distance of 3 m is set in front of the patient. With the start command, the patient gets up from his seat and walks 3 m, turns around and walks back and sits. With the start command, the time until the moment of sitting on the chair is recorded in seconds.Shorter duration indicates better functional mobility.
5 Times Sit To Stand Test(5XSST) | eight weeks
  5XSST evaluates lower extremity functional strength, transitional movements, balance and fall risk. The time it takes for the participant to sit and get up from a chair 5 times is recorded in seconds. Interpretations are made about balance and fall risk by comparing the norm times for age with the time the individual completes the test.
Cognitive Reserve Index Questionaire(CRIq) | eight weeks
  CRIq assesses an individual's cognitive reserve through compiling information about their entire adult life. If the participant has a suspected or confirmed cognitive weakness, the questionnaire must be answered by a family member or caregiver. The total score is obtained by recording the frequency of the individual's educational life, work and leisure activities in years. According to the score, the participant's cognitive reserve is interpreted as low, low - medium, medium, medium - high or high
Quality of Life in Alzheimer's Disease(QOL-AD) | eight weeks
  There are two versions of the scale: patient and family member/caregiver. In order to maximize construct validity, the scale is filled in independently by both patients and caregivers. It consists of questions asked about different aspects of life in order to determine the quality of life of the person. For each question, they are asked to choose the most appropriate one from the Poor, Fair, Good or Excellent answers.Higher scores indicate better quality of life.
Geriatric Depression Scale(GDS) | eight weeks
  The scale consists of 30 questions questioning how the participant felt in the past week. The person is asked to give the appropriate Yes(0) or No(1) answer to each question.Scores higher than 5 indicate depression.

SECONDARY OUTCOMES:
Dual-Task Questionnaire(DTQ) | eight weeks
  The Dual Task Questionnaire assesses the frequency of difficulties experienced by individuals with neurological injury or disease during activities of daily living that involve dual tasks. DTQ is scored between 0-40. Higher scores indicate more frequent dual-task difficulties.
Modified Falling Efficacy Scale(MFES) | eight weeks
  The scale consists of 14 items. On a scale of 0 to 10 (on the scale), the participant asked how safe they feel doing each of these activities without falling, with 0 being "not safe/not sure", 5 "quite safe/quite confident", and 10 "completely safe/ are asked to rate it in terms of being completely sure.
Mini Mental Test(MMT) | eight weeks
  Scoring is made between 0-30 on the scale in which the sub-headings of orientation, recording memory, attention and calculation, recall, language are evaluated.Lesser scores indicate worse cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Sevnaz ŞAHIN, PhD, Study Chair — Ege University
Locations (1):
- Karsiyaka Municipality Day Living Center, Izmir, Karsıyaka, Turkey (Türkiye)